CLINICAL TRIAL: NCT05243953
Title: Hypersensitivity to Opening of ATP-Sensitive Potassium Channels in Post-Traumatic Headache: A Randomized Clinical Trial
Brief Title: Hypersensitivity to Opening of ATP-Sensitive Potassium Channels in Post-Traumatic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Håkan Ashina, MD, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-21043704
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Post-Traumatic Headache
Keywords: Headache; Pain
MeSH Terms: conditions — Post-Traumatic Headache; Headache; Pain | interventions — Cromakalim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Experimental): A time- and volume-controlled infusion pump is used to administer levcromakalim by intravenous infusion over 20 minutes.
  Interventions: Drug: Levcromakalim
- Placebo (isotonic saline) (Placebo Comparator): A time- and volume-controlled infusion pump is used to administer placebo (isotonic saline) by intravenous infusion over 20 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levcromakalim — Study participants will be allocated to receive continuous intravenous infusion of 0.05 mg/min (20 ml of 50 mg/ml) levcromakalim.
  Arms: Levcromakalim
Drug: Placebo — Study participants will be allocated to receive continuous intravenous infusion of 20 mL placebo (isotonic saline).
  Other Names: Isotonic Saline
  Arms: Placebo (isotonic saline)

SUMMARY:
The aim is to investigate whether opening of ATP-sensitive potassium (KATP) channels induces headache with migraine-like features in people with persistent post-traumatic headache (PTH) attributed to mild traumatic brain injury (mTBI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* History of persistent headache attributed to mild traumatic injury to the head for ≥ 12 months and in accordance with the International Classification of Headache Disorders, 3rd Edition (ICHD-3)
* ≥ 4 monthly headache days on average across the 3 months prior to screening
* Provision of informed consent prior to initiation of any study-specific activities/procedures.

Exclusion Criteria:

* > 1 mild traumatic injury to the head
* History of any primary or secondary headache disorder prior to mild traumatic injury to the head (except for infrequent episodic tension-type headache)
* History of moderate or severe injury to the head
* History of whiplash injury
* History of craniotomy
* History or evidence of any other clinically significant disorder, condition or disease (except for those outlined above) than, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Initiation, discontinuation, or change of dosing of prophylactic medications within 2 months prior to study inclusion
* Intake of acute medications (e.g. analgesics, triptans) within 48 hours of infusion start
* Baseline headache intensity of >3 on an 11-point numeric rating scale (0 being no headache, 10 being the worst imaginable headache)
* Baseline headache with migraine-like features or self-reported baseline headache that mimics the subjects' usual headache with migraine-like features

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Migraine-Like Headache | 12 Hours
  Difference in incidence of headache with migraine-like features (0 to 12 hours) between levcromakalim and placebo.

SECONDARY OUTCOMES:
Headache Intensity Scores | 12 Hours
  Difference in area under the curve (AUC) for headache intensity scores (0 to 12 hours) between levcromakalim and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Ashina, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Denmark

REFERENCES:
- [Derived] Al-Khazali HM, Christensen RH, Dodick DW, Chaudhry BA, Burstein R, Ashina H. Hypersensitivity to opening of ATP-sensitive potassium channels in post-traumatic headache. Cephalalgia. 2023 Nov;43(11):3331024231210930. doi: 10.1177/03331024231210930. PMID 37917826